CLINICAL TRIAL: NCT06987513
Title: RECLAIM STUDY: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled Study Evaluating the Efficacy and Safety of Pemvidutide in the Treatment of Alcohol Use Disorder (AUD) in Subjects With Obesity or Overweight
Brief Title: RECLAIM STUDY: A Phase 2 Evaluating the Efficacy and Safety of Pemvidutide in the Treatment of Alcohol Use Disorder (AUD) in Subjects With Obesity or Overweight
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Altimmune, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALT-801-231
Record Dates: First submitted 2025-05-16; First posted 2025-05-23 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Alcohol Use Disorder (AUD)
Keywords: Pemvidutide; GLP-1 receptor agonist; Alcohol Use Disorder; Obesity; Overweight; AUD treatment; Phase 2
MeSH Terms: conditions — Alcoholism; Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pemvidutide 2.4mg (Active) (Experimental): Subcutaneous injection
  Interventions: Drug: Pemvidutide
- Placebo (Placebo Comparator): Subcutaneous injection
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Pemvidutide — Pemvidutide 2.4mg
  Arms: Pemvidutide 2.4mg (Active)
Other: Placebo — Subcutaneous injection
  Arms: Placebo

SUMMARY:
This is a Phase 2, multicenter, randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of pemvidutide in the treatment of AUD in subjects with obesity or overweight. After signing the informed consent form, subjects will be screened and if eligible randomized 1:1 to 1 of the following 2 treatment arms:

* Pemvidutide: 2.4 mg SC once weekly
* Placebo: Placebo SC once weekly

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent signed prior to performance of any study procedures
2. Male or female ages 18 to 75 years, inclusive
3. Diagnosis of current AUD of moderate or greater severity according to DSM-5 criteria
4. Reported drinking at least 28 drinks per week if male or 21 drinks per week if female in the 28 days prior to signing the informed consent. This should include at least 3 heavy drinking days per week (defined as ≥ 5 drinks per day for men and ≥ 4 drinks per day for women) Note: Baseline heavy drinking days will be determined by the TFLB method (28-day recall) drinking pattern collected at the initial screening visit
5. Overweight or obesity, defined as BMI ≥ 25 kg/m2

Exclusion Criteria:

1. Presence of clinically significant alcohol withdrawal symptoms, as defined as CIWA-Ar score ≥ 10 at screening and/or prior to randomization
2. History of hospitalization for alcohol intoxication or alcohol withdrawal
3. History of alcohol-related disorders including seizures related to alcohol, MalloryWeiss Syndrome, and alcoholic ketoacidosis
4. History and/or current DSM-5 diagnosis of schizophrenia, bipolar disorder, psychotic disorder or other severe psychiatric disorders, unless documented as well-controlled by the Investigator and cleared by the Medical Monitor
5. C-SSRS score indicative of active suicidal thoughts (answering "yes" to any of Questions 2 through 5 on the C-SSRS) in the past 6 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2025-05-15 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the average number of heavy drinking days per week, with a heavy drinking day defined as 5 or more drinks in the day for men and 4 or more drinks in the day for women, using the TLFB method | Week 24

SECONDARY OUTCOMES:
Proportion of subjects achieving a 2-level reduction in WHO risk drinking level using the TLFB method for the 4-week period comprising Weeks 21 through 24. | Week 24
Absolute change from baseline in average phosphatidylethanol (PEth) levels at Week 24 | 24 Weeks

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Altimmune Clinical Study Site, Los Angeles, California
  - Altimmune Clinical Study Site, Aurora, Colorado
  - Altimmune Clinical Study Site, New Haven, Connecticut
  - Altimmune Clinical Study Site, Fort Myers, Florida
  - Altimmune Clinical Study Site, University Park, Florida
  - Altimmune Clinical Study Site, North Canton, Ohio
  - Altimmune Clinical Study Site, Tulsa, Oklahoma
  - Altimmune Clinical Study Site, Philadelphia, Pennsylvania
  - Altimmune Clinical Study Site, Providence, Rhode Island
  - Altimmune Clinical Study Site, Charleston, South Carolina
  - Altimmune Clinical Study Site, Charlottesville, Virginia
  - Altimmune Clinical Study Site, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
It is anticipated that the results of this study will be presented at scientific meetings and/or published in a peer reviewed scientific or medical journal. A Publications Committee, comprised of the Investigators participating in the study and representatives from the Sponsor, as appropriate, will be formed to oversee the publication of the study results, which will reflect the experience of all participating study centers. Subsequently, individual Investigators may publish results from the study in compliance with their agreement with the Sponsor.